CLINICAL TRIAL: NCT03636503
Title: A Multi-Cohort Phase 1b Clinical Trial of Rituximab in Combination With Immunotherapy in Untreated and Previously Treated Follicular Lymphoma
Brief Title: Rituximab + Immunotherapy in Follicular Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Stopped was stopped prematurely due to drug manufacturer withdrawing supply/funding. Patients already enrolled on study were allowed to continue treatment.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Caron A. Jacobson, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-311
Record Dates: First submitted 2018-08-02; First posted 2018-08-17 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Follicular Lymphoma
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma | interventions — Rituximab; utomilumab; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Rituximab+Utomilumab+Avelumab-3mg (Experimental): * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * Utomilumab is administered intravenously over 1 hour once every 4 weeks
  * Avelumab is administered intravenously over 1 hour once every 2 weeks, 3mg/kg
  Interventions: Drug: Rituximab; Drug: Utomilumab; Drug: Avelumab
- Rituximab+Utomilumab+Avelumab-10mg (Experimental): * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * Utomilumab is administered intravenously over 1 hour once every 4 weeks
  * Avelumab is administered intravenously over 1 hour once every 2 weeks, 10mg/kg
  Interventions: Drug: Rituximab; Drug: Utomilumab; Drug: Avelumab
- PF04518600-0.3mg (Experimental): -PF-04518600 is administered intravenously over 1 hour on day 1 and day 15, 0.3mg/kg
  Interventions: Drug: PF04518600
- Rituximab+PF04518600-0.3mg (Experimental): * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * PF-04518600 is administered intravenously over 1 hour on day 1 and day 15, 0.3mg/kg
  Interventions: Drug: Rituximab; Drug: PF04518600
- Rituximab+Utomilumab+PF04518600-0.3mg (Experimental): * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * Utomilumab is administered intravenously over 1 hour once every 4 weeks
  * PF-04518600 is administered intravenously over 1 hour on day 1 and day 15, 0.3mg/kg
  Interventions: Drug: Rituximab; Drug: Utomilumab; Drug: PF04518600
- Rituximab+PF04518600-0.3mg+Avelumab-3mg (Experimental): * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * Utomilumab is administered intravenously over 1 hour once every 4 weeks
  * Avelumab is administered intravenously over 1 hour once every 2 weeks, 3mg/kg
  Interventions: Drug: Rituximab; Drug: Avelumab; Drug: PF04518600
- Rituximab+PF04518600-0.3mg+Avelumab-10mg (Experimental): * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * Utomilumab is administered intravenously over 1 hour once every 4 weeks
  * Avelumab is administered intravenously over 1 hour once every 2 weeks, 10mg/kg
  Interventions: Drug: Rituximab; Drug: Avelumab; Drug: PF04518600

INTERVENTIONS:
Drug: Rituximab — Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  Other Names: Rituxan
  Arms: Rituximab+PF04518600-0.3mg; Rituximab+PF04518600-0.3mg+Avelumab-10mg; Rituximab+PF04518600-0.3mg+Avelumab-3mg; Rituximab+Utomilumab+Avelumab-10mg; Rituximab+Utomilumab+Avelumab-3mg; Rituximab+Utomilumab+PF04518600-0.3mg
Drug: Utomilumab — Utomilumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  Other Names: PF-05082566; PF05082566
  Arms: Rituximab+Utomilumab+Avelumab-10mg; Rituximab+Utomilumab+Avelumab-3mg; Rituximab+Utomilumab+PF04518600-0.3mg
Drug: Avelumab — Avelumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  Other Names: Bavencio
  Arms: Rituximab+PF04518600-0.3mg+Avelumab-10mg; Rituximab+PF04518600-0.3mg+Avelumab-3mg; Rituximab+Utomilumab+Avelumab-10mg; Rituximab+Utomilumab+Avelumab-3mg
Drug: PF04518600 — In the presence of tumor-associated antigens (TAAs), this may promote a T-cell-mediated immune response against TAA-expressing tumor cells. OX40
  Other Names: PF-04518600
  Arms: PF04518600-0.3mg; Rituximab+PF04518600-0.3mg; Rituximab+PF04518600-0.3mg+Avelumab-10mg; Rituximab+PF04518600-0.3mg+Avelumab-3mg; Rituximab+Utomilumab+PF04518600-0.3mg

SUMMARY:
This research study is studying several new investigational drug combinations as a possible treatment for follicular lymphoma.

The drugs involved are:

* Rituximab
* Utomilumab
* Avelumab
* PF-04518600

DETAILED DESCRIPTION:
This research study is a Phase 1 clinical trial. Phase 1 clinical trials test the safety of an investigational intervention and also try to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

Utomilumab and avelumab are drugs which may stimulate the immune system against tumor cells. Because they activate the immune system, they are sometimes called immunotherapy drugs. The FDA (the U.S. Food and Drug Administration) has not approved utomilumab or avelumab for treatment of this cancer.

Rituximab is approved by the FDA (the U.S. Food and Drug Administration) as a treatment option for this disease.

The purpose of this research is to learn about the effects of combining the immunotherapy drugs utomilumab and avelumab with rituximab in follicular lymphoma. The investigators hope to learn how safe the combinations of treatments are for participants with follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically determined follicular lymphoma, grade 1-3A, with pathologic review at the participating institutions, that has either:

  * Relapsed or primary refractory after at least one line of therapy including anti-CD-20 monoclonal antibody treatment (part A) or;
  * Has had no previous anti-lymphoma therapy other than corticosteroids or radiotherapy (part B).
* Patients with active histologic transformation are excluded. Relapsed/refractory patients with prior transformation may be included as long as there is no evidence of transformation at the time of study entry by pathology, imaging, or clinical status
* Patients in part B, without prior anti-lymphoma therapy, must be in need of treatment as defined by any of the following criteria:

  * Symptomatic adenopathy
  * Organ function impairment due to disease involvement, including cytopenias due to marrow involvement (WBC <1.5x109/L; absolute neutrophil count [ANC] <1.0x109/L, Hgb <10g/dL; platelets <100x109/L)
  * Constitutional symptoms
  * Maximum diameter of disease > 7cm

    -->3 nodal sites of involvement
  * Risk of local compressive symptoms
  * Splenomegaly (craniocaudal diameter > 16cm on CT imaging)
  * Clinically significant pleural or peritoneal effusion
  * Leukemic phase (>5x109/L circulating malignant cells)
  * Rapid generalized disease progression
  * Renal infiltration
  * Bone lesions
* Patients may have had a prior autologous stem cell transplant and may have been treated with autologous chimeric antigen receptor T-cells (CAR T-cells).
* Not in need of urgent cytoreductive therapy in the opinion of the investigator
* Measurable disease that has not been previously irradiated on CT scans of at least 1.5 cm, OR if the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation. Imaging must be completed no greater than 6 weeks prior to study enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (see Appendix A)
* Adequate hematologic and organ function:

  * Absolute neutrophil count > 1.0x109/L unless due to marrow involvement by lymphoma in which case ANC must be >0.5x109/L
  * Platelets > 75 x109/L, unless due to marrow involvement by lymphoma, in which case platelets must be >50 x109/L
  * Creatinine < 1.5 x ULN (upper limit of normal) or estimated GFR > 40ml/min
  * Total bilirubin < 1.5 X ULN, unless Gilbert syndrome, in which case direct bilirubin must be < 3 x ULN
* AST/ALT < 2.5 X ULN, unless documented liver involvement by lymphoma, in which case AST/ALT must be <5 x ULN
* Age >18 years
* Ability to understand and the willingness to sign a written informed consent document.
* Willingness to provide pre-treatment (or recent archival w/o intervening therapy), and on-treatment tumor samples by core needle or excisional surgical biopsy

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 28 days of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc.), or 56 days for radioimmunotherapy. Steroids for symptom palliation are allowed, but must be either discontinued or on stable doses of < 10mg daily of prednisone (or the equivalent) at the time of initiation of protocol therapy.
* Patients may not be receiving any other investigational agents, or have received investigational agents within 4 weeks (or 3 half-lives, whichever is longer) of beginning treatment.
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy unless in consultation with an allergy specialist they are deemed eligible for retreatment with desensitization.
* Patients who have previously received therapy with any drug that works by a similar mechanism of action as any drug being tested in a given cohort will be excluded from that cohort but will be allowed to enroll in other open cohorts.
* Patients who have undergone prior allogeneic stem cell transplantation
* Patients with a history of or active autoimmune disease (except controlled asthma, Hashimoto thyroiditis, atopic dermatitis, and/or vitiligo), or requiring systemic corticosteroids at a dose of 10mg prednisone equivalent daily. Patients with a history of autoimmune disease who never required corticosteroids and with no evidence of disease activity, and in whom the risk of reactivation is felt not to be serious, may be enrolled after discussion with the overall study chair. Exceptions to this are patients with a history of inflammatory bowel disease (ulcerative colitis and Crohn's disease). These patients are excluded regardless of whether their disease is active or inactive.
* Patients with active pneumonitis or colitis, or patients with chronic liver disease and/or cirrhosis
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study.
* Patients with known leptomeningeal or brain metastases. Imaging or spinal fluid analysis to exclude CNS involvement is not required, unless there is clinical suspicion by the treating investigator.
* Patients with known HIV infection or hepatitis B or C infection. Testing for HIV is optional. Testing for hepatitis B and C is mandatory. Patients with hepatitis B core Ab positivity but negative surface antigen and negative viral load may be enrolled if they can be treated with a prophylactic agent (eg, entecavir); patients with hepatitis C seropositivity who have undergone successful treatment with negative viral load can also be enrolled.
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Prior history of another malignancy (except for non-melanoma skin cancer or in situ cervical or breast cancer) unless disease free for at least three years. Patients with prostate cancer are allowed if PSA is less than 1.
* Patients should not have received immunization with attenuated live vaccine within one week of study entry or during study period.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. Women of child bearing potential (WOCBP) or male study participants of reproductive potential must agree to use double barrier birth control method of contraception during the course of the study treatment period and for 3 months after completing study treatment. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who are not postmenopausal (no menses) for at least 12 consecutive months. WOCBP must have a negative urine or serum pregnancy test within 14 days prior to administration of treatment.
* History of noncompliance to medical regimens.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * New York Heart Association Class III or IV cardiac disease, including pre-existing clinically significant arrhythmia, congestive heart failure, or cardiomyopathy
  * Patients with a history of previous anthracycline treatment and are at risk of cardiac failure (New York Heart Association Class II or above) are excluded from cohorts A2, A3, and B2 (cohorts that include PF04518600)
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
* Patients with any one of the following currently on or in the previous 6 months will be excluded from cohorts A2, A3, and B2 (any cohort that includes treatment with PF04518600) myocardial infarction, congenital long QT syndrome, torsade's de points, left anterior hemiblock (bifascicular block), unstable angina, coronary/peripheral artery bypass graft, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism or other clinically significant episode of thrombo-embolic disease*. Ongoing cardiac dysrhythmias of NCI CTCAE grade > 2, atrial fibrillation of any grade, or QTcF interval >470msec at screening (except in case of right bundle branch block, these cases must be discussed with the principal investigator). *Cases must be discussed in detail with the principal investigator to judge eligibility. Anticoagulation (heparin only, no vitamin K antagonists or factor Xa inhibitors will be allowed if indicated.
* Other uncontrolled intercurrent illness that would limit adherence to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caron A. Jacobson, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (6):
- United States (6):
  - City of Hope, Duarte, California
  - Yale New-Haven Hospital, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merryman RW, Redd RA, Freedman AS, Ahn IE, Brown JR, Crombie JL, Davids MS, Fisher DC, Jacobsen ED, Kim AI, LaCasce AS, Ng S, Odejide OO, Parry EM, Isufi I, Kline J, Cohen JB, Mehta-Shah N, Bartlett NL, Mei M, Kuntz TM, Wolff J, Rodig SJ, Armand P, Jacobson CA. A multi-cohort phase 1b trial of rituximab in combination with immunotherapy doublets in relapsed/refractory follicular lymphoma. Ann Hematol. 2024 Jan;103(1):185-198. doi: 10.1007/s00277-023-05475-0. Epub 2023 Oct 18. PMID 37851072

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated early due to the drug manufacturer stopping drug supply.
Groups:
- Rituximab+Utomilumab+Avelumab-3mg: * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * Utomilumab is administered intravenously over 1 hour once every 4 weeks
  * Avelumab is administered intravenously over 1 hour once every 2 weeks, 3mg
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  Utomilumab: Utomilumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  Avelumab: Avelumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
- Rituximab+Utomilumab+Avelumab-10mg: * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * Utomilumab is administered intravenously over 1 hour once every 4 weeks
  * Avelumab is administered intravenously over 1 hour once every 2 weeks, 10mg
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  Utomilumab: Utomilumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  Avelumab: Avelumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
- Rituximab+PF04518600-0.3mg: * Rituximab is administered intravenously per institutional standards
  * PF-04518600 is administered intravenously over 1 hour on day 1 and day 15, 0.3mg/kg
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  PF04518600: In the presence of tumor-associated antigens (TAAs), this may promote a T-cell-mediated immune response against TAA-expressing tumor cells. OX40
- Rituximab+Utomilumab+PF04518600-0.3mg: * Rituximab is administered intravenously per institutional standards
  * Utomilumab is administered intravenously over 1 hour once every
  * PF-04518600 is administered intravenously over 1 hour on day 1 and day 15, 0.3mg/kg
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  Utomilumab: Utomilumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  PF04518600: In the presence of tumor-associated antigens (TAAs), this may promote a T-cell-mediated immune response against TAA-expressing tumor cells. OX40
- Rituximab+PF04518600-0.3mg+Avelumab-3mg: * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * Avelumab is administered intravenously over 1 hour once every 2 weeks, 3mg/kg
  * PF-04518600 is administered intravenously over 1 hour on day 1 and day 15, 0.3mg/kg
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  PF04518600: In the presence of tumor-associated antigens (TAAs), this may promote a T-cell-mediated immune response against TAA-expressing tumor cells. OX40
  Avelumab: Avelumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
- Rituximab+PF04518600-0.3mg+Avelumab-10mg: * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * PF-04518600 is administered intravenously over 1 hour on day 1 and day 15, 0.3mg/kg
  * Avelumab is administered intravenously over 1 hour once every 2 weeks, 10mg/kg
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  PF04518600: In the presence of tumor-associated antigens (TAAs), this may promote a T-cell-mediated immune response against TAA-expressing tumor cells. OX40
  Avelumab: Avelumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
Period: Overall Study
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Started | 5 | 4 | 3 | 3 | 9 | 0 | 0
Completed | 5 | 4 | 3 | 3 | 9 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of unique patients analyzed is 24; however, one patient was treated on two arms (Rituximab+Utomilumab+Avelumab-10mg and Rituximab+PF04518600-0.3mg)
Groups:
- Rituximab+Utomilumab+Avelumab-10mg: * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * Utomilumab is administered intravenously over 1 hour once every 4 weeks
  * Avelumab is administered intravenously over 1 hour once every 2 weeks, 10mg
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  Utomilumab: Utomilumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  Avelumab: Avelumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  -PF-04518600 is administered intravenously over 1 hour on day 1 and day 15, 0.3mg/kg
- Total: Total of all reporting groups
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg | Total
Number analyzed (Participants) | 5 | 4 | 3 | 3 | 9 | 0 | 0 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 2 | 1 | 7 | 0 | 0 | 17
  >=65 years | 0 | 2 | 1 | 2 | 2 | 0 | 0 | 7
Age, Continuous [Median (Full Range); unit: years] | 58 [51 to 62] | 61 [42 to 76] | 58 [50 to 72] | 65 [42 to 66] | 57 [46 to 76] |  |  | 58 [42 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 6
  Male | 5 | 2 | 3 | 1 | 7 | 0 | 0 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 4 | 3 | 3 | 8 | 0 | 0 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  White | 5 | 4 | 3 | 2 | 8 | 0 | 0 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 3 | 3 | 9 | 0 | 0 | 24
ECOG Performance Status [Count of Participants; unit: Participants]
  0 - Fully active, able to carry on all pre-disease performance without restriction | 1 | 2 | 1 | 2 | 6 | 0 | 0 | 12
  1 - Restricted in physically strenuous activity but able to carry out light or sedentary work | 4 | 2 | 2 | 1 | 3 | 0 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dosing
Description: Patients assessed for DLT after each 28-day cycle of treatment. Up to two cohorts of 3 patients per dose level plus expansion cohort.
  Rituximab/Utomilumab/Avelumab arm assessed 2 dose levels. Rituximab/Utomilumab/PF04518600 assessed 3 dose levels. Rituximab/PF04518600/Avelumab assessed 2 dose levels.
Time Frame: 6 months total, assessed after each 28-day cycle
Population: All patients treated with any amount of study treatment. One patient was included separately in arms 1 (Rituximab+Utomilumab+Avelumab-3mg) and 3 (PF04518600-0.3mg)
Measure: Number; unit: mg
Groups:
- Rituximab/Utomilumab/Avelumab - Level 1: Dose level 1: Rituximab 375mg/m2 IV q7 days x 4 doses, utomilumab 100mg IV q28d, avelumab 3mg/kg IV q14 days
  * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * Utomilumab is administered intravenously over 1 hour once every 4 weeks
  * Avelumab is administered intravenously over 1 hour once every 2 weeks
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  Utomilumab: Utomilumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  Avelumab: Avelumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
- Rituximab/Utomilumab/Avelumab - Level 2: Dose level 2: Rituximab 375mg/mg2 IV q7 days x 4 doses, utomilumab 100mg IV q28d, avelumab 10mg/kg IV q14 days
  * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * Utomilumab is administered intravenously over 1 hour once every 4 weeks
  * Avelumab is administered intravenously over 1 hour once every 2 weeks
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  Utomilumab: Utomilumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  Avelumab: Avelumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
- Rituximab/Utomilumab/PF04518600 - Level 1: Dose level 0: PF-04518600 0.3mg/kg IV q14 days
  * Rituximab is administered intravenously per institutional standards
  * Utomilumab is administered intravenously over 1 hour once every
  * PF-04518600 is administered intravenously over 1 hour on day 1 and day 15
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  Utomilumab: Utomilumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  PF04518600: In the presence of tumor-associated antigens (TAAs), this may promote a T-cell-mediated immune response against TAA-expressing tumor cells. OX40
- Rituximab/Utomilumab/PF04518600 - Level 2: Dose level 1: Rituximab 375mg/m2 IV q7 days x 4 doses, PF-04518600 0.3mg/kg IV q14 days
  * Rituximab is administered intravenously per institutional standards
  * Utomilumab is administered intravenously over 1 hour once every
  * PF-04518600 is administered intravenously over 1 hour on day 1 and day 15
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  Utomilumab: Utomilumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  PF04518600: In the presence of tumor-associated antigens (TAAs), this may promote a T-cell-mediated immune response against TAA-expressing tumor cells. OX40
- Rituximab/Utomilumab/PF04518600 - Level 3: Dose level 2: Rituximab 375mg/m2 IV q7 days x 4 doses, PF-04518600 0.3mg/kg IV q14 days, utomilumab 100mg IV q28 days
  * Rituximab is administered intravenously per institutional standards
  * Utomilumab is administered intravenously over 1 hour once every
  * PF-04518600 is administered intravenously over 1 hour on day 1 and day 15
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  Utomilumab: Utomilumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
  PF04518600: In the presence of tumor-associated antigens (TAAs), this may promote a T-cell-mediated immune response against TAA-expressing tumor cells. OX40
- Rituximab/PF04518600/Avelumab - Level 1: Dose level 1: Rituximab 375mg/m2 IV q7 days x 4 doses, PF-04518600 0.3mg/kg IV q14 days, avelumab 3mg/kg IV q14 days
  * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * PF-04518600 is administered intravenously over 1 hour on day 1 and day 15
  * Avelumab is administered intravenously over 1 hour once every 2 weeks
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  PF04518600: In the presence of tumor-associated antigens (TAAs), this may promote a T-cell-mediated immune response against TAA-expressing tumor cells. OX40
  Avelumab: Avelumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
- Rituximab/PF04518600/Avelumab - Level 2: Dose level 2: Rituximab 375mg/m2 IV q7 days x 4 doses, PF-04518600 0.3mg/kg IV q14 days, avelumab 10mg/kg IV q14 days
  * Rituximab is administered intravenously per institutional standards for four weekly treatments for cycle 1 only
  * PF-04518600 is administered intravenously over 1 hour on day 1 and day 15
  * Avelumab is administered intravenously over 1 hour once every 2 weeks
  Rituximab: Rituximab works by targeting the CD20 antigen on normal and malignant B-cells. Then the body's natural immune defenses are recruited to attack and kill the marked B-cells. Stem cells (young cells in the bone marrow that will develop into the various types of cells) do not have the CD20 antigen. This allows healthy B-cells to regenerate after treatment
  PF04518600: In the presence of tumor-associated antigens (TAAs), this may promote a T-cell-mediated immune response against TAA-expressing tumor cells. OX40
  Avelumab: Avelumab is a drug which may stimulate the immune system against tumor cells. Because it activate the immune system, it is sometimes called immunotherapy drug
Arm/Group | Rituximab/Utomilumab/Avelumab - Level 1 | Rituximab/Utomilumab/Avelumab - Level 2 | Rituximab/Utomilumab/PF04518600 - Level 1 | Rituximab/Utomilumab/PF04518600 - Level 2 | Rituximab/Utomilumab/PF04518600 - Level 3 | Rituximab/PF04518600/Avelumab - Level 1 | Rituximab/PF04518600/Avelumab - Level 2
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
mg
  Rituximab | 375 | 375 | NA — This cohort did not receive this treatment | 375 | 375 |  |
  PF-04518600 | NA — This cohort did not receive this treatment | NA — This cohort did not receive this treatment | 0.3 | 0.3 | 0.3 |  |
  Utomilumab | 100 | 100 | NA — This cohort did not receive this treatment | NA — This cohort did not receive this treatment | 100 |  |
  Avelumab | 3 | 10 | NA — This cohort did not receive this treatment | NA — This cohort did not receive this treatment | NA — This cohort did not receive this treatment |  |

2. Primary Outcome: Number of Participants With Complete Response Per Lugano Criteria
Description: Per 2014 Lugano criteria, a complete response is defined as
  PET-CT, score 1, 2, or 3* with or without a residual mass on 5PS Or on CT, target nodes/nodal masses must regress to ≤ 1.5 cm in LDi, and no extralymphatic sites of disease
Time Frame: Response assessed after completing treatment (6 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
Participants | 0 | 1 | 0 | 0 | 2 |  |

3. Secondary Outcome: Number of Participants With Partial Response Per Lugano Criteria
Description: Per 2014 Lugano criteria, partial response is defined as
  PET-CT Score 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size Or On CT ≥ 50% decrease in SPD of up to 6 target measurable nodes and extranodal sites; no increase in non-measured lesions; spleen if enlarged must have regressed by >50% in length beyond normal
Time Frame: Response assessed after completing treatment (6 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
Participants | 2 | 1 | 0 | 0 | 1 |  |

4. Secondary Outcome: Number of Participants With Objective Response Per Lugano Criteria
Description: Objective response rate is defined as complete + partial response (CR + PR)
  Per 2014 Lugano criteria, CR is defined as
  PET-CT, score 1, 2, or 3* with or without a residual mass on 5PS Or on CT, target nodes/nodal masses must regress to ≤ 1.5 cm in LDi, and no extralymphatic sites of disease
  Per 2014 Lugano criteria, PR is defined as
  PET-CT Score 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size.
  Or On CT ≥ 50% decrease in SPD of up to 6 target measurable nodes and extranodal sites; no increase in non-measured lesions; spleen if enlarged must have regressed by >50% in length beyond normal
Time Frame: Response assessed after completing treatment (6 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
Participants | 2 | 2 | 0 | 0 | 3 |  |

5. Secondary Outcome: Number of Participants With Objective Response Per LYRIC Criteria
Description: Objective response rate is defined as complete + partial response (CR + PR)
  Per LYRIC criteria, CR is defined as
  PET-CT, score 1, 2, or 3* with or without a residual mass on 5PS Or on CT, target nodes/nodal masses must regress to ≤ 1.5 cm in LDi, and no extralymphatic sites of disease
  Per LYRIC criteria, PR is defined as
  PET-CT Score 4 or 5 with reduced uptake compared with baseline and residual mass(es) of any size.
  Or On CT ≥ 50% decrease in SPD of up to 6 target measurable nodes and extranodal sites; no increase in non-measured lesions; spleen if enlarged must have regressed by >50% in length beyond normal
Time Frame: Response assessed after completing treatment (6 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
Participants | 2 | 2 | 0 | 0 | 3 |  |

6. Secondary Outcome: Number of Participants With Complete Response Per LYRIC Criteria
Description: Per LYRIC criteria, complete response is defined as
  PET-CT, score 1, 2, or 3* with or without a residual mass on 5PS Or on CT, target nodes/nodal masses must regress to ≤ 1.5 cm in LDi, and no extralymphatic sites of disease
Time Frame: Response assessed after completing treatment (6 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
Participants | 0 | 1 | 0 | 0 | 2 |  |

7. Secondary Outcome: Progression-Free Survival Per Lugano Criteria
Description: Time from registration until earlier of progression (Lugano criteria) or death from any cause, censored at date last known alive and progression-free
Time Frame: 6 cycles (approximately 6 months) of treatment followed by 24 months of active follow-up with contact every 3 months
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
months | 7.0 [0 to 12.6] | 6.1 [3.0 to 7.5] | 2.7 [1.5 to 12.7] | 2.4 [0.0 to 3.2] | 6.8 [0.0 to 12.5] |  |

8. Secondary Outcome: Progression-Free Survival Per LYRIC Criteria
Description: Time from registration until earlier of progression (LYRIC criteria) or death from any cause, censored at date last known alive and progression-free
Time Frame: 6 cycles (approximately 6 months) of treatment followed by 24 months of active follow-up with contact every 3 months
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
months | 7.2 [0 to 12.6] | 6.1 [3.0 to 7.5] | 2.7 [1.5 to 12.7] | 2.4 [0.0 to 3.2] | NA [0.0 to 12.5] — The median PFS has not yet been reached |  |

9. Secondary Outcome: Overall Survival
Description: Time from registration until death from any cause, censored at date last known alive
Time Frame: 6 cycles (approximately 6 months) of treatment followed by 24 months of active follow-up with contact every 3 months followed by 3-year survival follow-up with contact every 6 months
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
months | 28.2 [14.1 to 36.3] | 12.9 [2.3 to 19.0] | NA [31.8 to 36.7] — The median OS has not yet been reached due to an insufficient number of events. No deaths were observed in this cohort--full ranges include censoring/follow-up times. | NA [0.3 to 16.9] — The median OS has not yet been reached due to an insufficient number of events. No deaths were observed in this cohort--full ranges include censoring/follow-up times. | NA [2.2 to 15.6] — The median OS has not yet been reached due to an insufficient number of events. No deaths were observed in this cohort--full ranges include censoring/follow-up times. |  |

10. Secondary Outcome: Number of Participants With Grade 3 and Higher Toxicities
Description: Number of patients who experience any adverse event with grade 3 or higher regardless of attribution to one or more study treatments
Time Frame: 6 cycles (approximately 6 months) of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
Participants | 5 | 2 | 0 | 2 | 2 |  |

11. Secondary Outcome: Number of Participants With Grade 3 and Higher Related Toxicities
Description: Number of patients who experience any adverse event with grade 3 or higher related to one or more study treatments
Time Frame: 6 cycles (approximately 6 months) of treatment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
Participants | 3 | 0 | 0 | 2 | 2 |  |

12. Secondary Outcome: Number of Participants With Grade 2 or Higher Toxicity
Description: Number of patients who experience any adverse event with grade 2 or higher regardless of treatment attribution
Time Frame: 6 cycles (approximately 6 months) of treatment followed
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
Number analyzed (Participants) | 6 | 4 | 3 | 3 | 9 | 0 | 0
Participants | 6 | 3 | 0 | 3 | 8 |  |

ADVERSE EVENTS:
Time Frame: Adverse events collected starting at baseline over each of 6 cycles of treatment (for 28-day cycles) and up to 30 days after last dose of treatment or until resolution of toxicity to grade 1 or baseline. All-Cause Mortality was monitored up to 4 years (6 cycles (approximately 6 months) of treatment followed by 24 months of active follow-up with contact every 3 months followed by 3-year survival follow-up with contact every 6 months).
Description: There were no patients treated on arm 3, Rituximab+Avelumab+PF04518600. One patient was included separately in arms 1 (Rituximab+Utomilumab+Avelumab-3mg) and 3 (PF04518600-0.3mg).
Arm/Group | Rituximab+Utomilumab+Avelumab-3mg | Rituximab+Utomilumab+Avelumab-10mg | PF04518600-0.3mg | Rituximab+PF04518600-0.3mg | Rituximab+Utomilumab+PF04518600-0.3mg | Rituximab+PF04518600-0.3mg+Avelumab-3mg | Rituximab+PF04518600-0.3mg+Avelumab-10mg
All-Cause Mortality (participants affected / at risk) | 2/6 | 1/4 | 0/3 | 0/3 | 0/9 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/6 | 0/4 | 0/3 | 1/3 | 1/9 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/6 | 3/4 | 2/3 | 3/3 | 6/9 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab+Utomilumab+Avelumab-3mg (N=6) | Rituximab+Utomilumab+Avelumab-10mg (N=4) | PF04518600-0.3mg (N=3) | Rituximab+PF04518600-0.3mg (N=3) | Rituximab+Utomilumab+PF04518600-0.3mg (N=9) | Rituximab+PF04518600-0.3mg+Avelumab-3mg (N=0) | Rituximab+PF04518600-0.3mg+Avelumab-10mg (N=0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — COVID-19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab+Utomilumab+Avelumab-3mg (N=6) | Rituximab+Utomilumab+Avelumab-10mg (N=4) | PF04518600-0.3mg (N=3) | Rituximab+PF04518600-0.3mg (N=3) | Rituximab+Utomilumab+PF04518600-0.3mg (N=9) | Rituximab+PF04518600-0.3mg+Avelumab-3mg (N=0) | Rituximab+PF04518600-0.3mg+Avelumab-10mg (N=0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Increased Lymphadenopathy
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — General Discomfort
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This trial was terminated early due to drug manufacturer discontinuing drug and no longer supplying.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT03636503/Prot_SAP_000.pdf